CLINICAL TRIAL: NCT06670547
Title: Prospective and Multicenter Spanish Registry of Quality Indicators and Adverse Events of Endoscopic Retrograde Cholangiopancreatography
Brief Title: Spanish Registry of Quality Indicators and Adverse Events of Endoscopic Retrograde Cholangiopancreatography
Status: Not yet recruiting | Type: Observational
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Spanish Society of Digestive Endoscopy (Other)
Responsible Party: Sponsor
Other Study IDs: PI-23-281
Record Dates: First submitted 2024-10-22; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Choledocholithiasis; Choledocholithiasis With Acute Cholangitis; Cholangiocarcinoma; Sclerosing Cholangitis; Pancreatic Cancer Resectable; Pancreatic Cancer Non-resectable; Biliary Fistula
Keywords: ERCP ADVERSE EVENTS; PERFORMANCE MEASURES
MeSH Terms: conditions — Choledocholithiasis; Cholangiocarcinoma; Cholangitis, Sclerosing; Biliary Fistula | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with biliopancreatic pathology undergoing ERCP: Patients with biliopancreatic pathology who undergo ERCP are over 18 years of age and sign the informed consent.
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography (ERCP)

INTERVENTIONS:
Procedure: Endoscopic retrograde cholangiopancreatography (ERCP) — Endoscopic retrograde cholangiopancreatography (ERCP)

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is a technique which combines endoscopic and radiological vision and allows for therapeutic procedures on pathologies of the pancreas and bile duct.

ERCP is a generally well tolerated procedure, nonetheless it is a complex technique that has a higher frequency of complications compared to most endoscopic procedures that can even be life-threatening. These complications are related to patient characteristics, experience of the endoscopist performing the procedure, and specific factors to the technique. Due to its complexity, quality assurance, operator training and auditing are required to increase success and minimize complications.

There are quality indicators suggested by the main scientific societies in relation to technical aspects and complications, recommending their monitoring and auditing. Most endoscopy units lack records to monitor quality and complications, which prevents the assessment of quality and the identification of areas for improvement.

Given the lack of evidence of the quality of ERCP in the Spanish population, the investigators will be conducting a multicenter, national prospective study that will include subjects who undergo ERCP.

Patient data and technical aspects of the procedure will be recorded and all included patients will be monitored to identify complications. The quality indicators obtained within the registry will be compared with those established by scientific societies and the relationship between complications and technical factors will be analyzed.

DETAILED DESCRIPTION:
Currently, endoscopic retrograde cholangiopancreatography (ERCP) is a well-established procedure that is in continuous development, with an incidence and severity of adverse events (AEs) that differ substantially from those related to other endoscopic procedures, reaching up to 14.7% and with a mortality rate of 0.7%, even in expert centers 1. For this reason, it is essential to ensure the quality of ERCP procedures, requiring optimal training, capacity building and auditing to increase the success of the procedure and minimize the risk of complications 2.

In recent years, the evaluation of the quality of ERCP has gained interest among health professionals and patient organizations. In 2018, the European Society of Gastrointestinal Endoscopy (ESGE) and the United European Gastroenterology (UEG) published key quality recommendations for ERCP and endoscopic ultrasonography with the aim of encouraging healthcare professionals to implement these performance targets at national level 3. For ERCP there are 5 recommendations including adequate antibiotic prophylaxis before ERCP (at least 90%), biliary cannulation rate (at least 90%), adequate stent placement in patients with sub-hilum obstruction (at least 95%), removal of bile duct stones (at least 90%) and post-ERCP pancreatitis (less than 10%).

Following this line, endoscopists in the Netherlands have been using a mandatory nationwide quality register since 2016 (Trans.IT database; Rotterdam, the Netherlands), which provides information on the quality of ERCP 4. They have recently published the analysis of this register in relation to the ESGE quality recommendations. 5671 procedures performed by 57 endoscopists in 11 centres were included. Three key quality indicators were met: successful biliary cannulation, adequate placement of stents for biliary obstruction and removal of bile duct stones with a high overall success rate. These robust data from routine clinical practice also allow us to identify areas for improving the quality of ERCP, for example, successful cannulation of native papillae below 90% for endoscopists performing fewer than 50 procedures per year or the rate of adequate placement of biliary stents below 90% in endoscopists performing fewer than 25 procedures per year 5. Unfortunately, the rate of pancreatitis, which is the most appropriate indicator of the rate of adverse events, was not evaluated in this registry.

In our view, the collection of data at a national level is of undoubted value to identify areas for improvement and to guarantee quality in ERCP, however, there are no state databases in our setting.

The present study aims to evaluate the quality indicators of ERCP recommended by the ESGE-UEG in a Spanish prospective registry and to describe the real incidence of adverse events in clinical practice, and their association with technical aspects of the procedure.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients who have undergone an ERCP at participating centres from 1 November 2024 will be included. An ERCP will be considered to have been performed when an endoscope is introduced to access the duodenal papilla.

These included patients must meet all of the following criteria:

* Over 18 years of age
* Signed informed consent.

Exclusion Criteria:

* Under 18 years of age
* Unavailability of informed consent
* Impossibility of follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biliopancreatic pathology for whom ERCP is performed in hospitals in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate compliance with ESGE-UEG ERCP quality indicators in the Spanish registry | Patients receiving antibiotic prophylaxis of at least one dose of any systemic antibiotic in a 12-hour interval prior to ERCP.
  Number of participants receiving adequate antibiotic prophylaxis before ERCP.
To evaluate compliance with ESGE-UEG ERCP quality indicators in the Spanish registry. | Patients in whom biliary cannulation is achieved up to 1 hour after completion of ERCP.
  Number of participants who achieved biliary cannulation.
To evaluate compliance with ESGE-UEG ERCP quality indicators in the Spanish registry. | Patients who successfully placed stents in obstructions distal to the hilum up to 1 hour after completion of ERCP.
  Number of participants in whom stents are successfully placed in obstructions distal to the hilum.
To evaluate compliance with ESGE-UEG ERCP quality indicators in the Spanish registry. | Patients who successfully removed bile duct stones up to 1 hour after completion of ERCP.
  Number of participants with successful removal of biliary tract stones.
To evaluate compliance with ESGE-UEG ERCP quality indicators in the Spanish registry. | Patients who developed acute pancreatitis at 7 and 30 days after ERCP.
  Number of participants developing post-ERCP pancreatitis.

SECONDARY OUTCOMES:
To describe the severity of adverse events in ERCP according to the AGREE classification and their association with technical aspects of the procedure | Assessment of the development of adverse events at 24 hours according to the practice of each hospital; at 7 days and at 30 days after performing the ERCP by telephone call.
  Number adverse event (AE)A telephone contact with general practitioner, outpatient clinic, or endoscopy service without any intervention or extended observation of the patient after the procedure (3 hours without any intervention)
  Grade I AE with any deviation of the standard post-procedural course, without pharmacologic treatment or endoscopic, radiologic, or surgical interventions, Hospital admission (24 hours), without any intervention, Allowed therapeutic regimens are antiemetics, antipyretics, analgesics and electrolytes or Allowed diagnostic radiology and laboratory tests
  Grade II AE requiring pharmacologic treatment with drugs other than those allowed for grade I AE or Blood product transfusions or Hospital admission for more than 24 hours
  Grade Illa AE requiring endoscopic or radiologic intervention Grade Illb Surgical intervention
  Grade IV AE requiring intensive care unit IVa Single-organ dysfunction including dialysis IVb Multiorgan dysfunction Grade V Death of patient

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Castillo-Regalado, MD, Principal Investigator — Hospital Universitario Germans Trias i Pujol (Badalona)

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in ERCP and biliopancreatic diseases. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
  Data requests can be submitted starting 10 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 10 months and ending 2 years after the publication of results.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement.

REFERENCES:
- [Background] Ministerio de Sanidad. Criterios homologados, acordados por el Consejo Interterritorial, que deben cumplir los CSUR para ser designados como de referencia del Sistema Nacional de Salud. Drenaje guiado por ecoendoscopia de la obstrucción biliopancreática compleja.
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Nass KJ, Zwager LW, van der Vlugt M, Dekker E, Bossuyt PMM, Ravindran S, Thomas-Gibson S, Fockens P. Novel classification for adverse events in GI endoscopy: the AGREE classification. Gastrointest Endosc. 2022 Jun;95(6):1078-1085.e8. doi: 10.1016/j.gie.2021.11.038. Epub 2021 Dec 8. PMID 34890695
- [Background] Brindise EM, Gerke H. Monitoring adverse events after ERCP: Call me maybe? Gastrointest Endosc. 2021 Apr;93(4):911-913. doi: 10.1016/j.gie.2020.08.036. No abstract available. PMID 33741091
- [Background] Theunissen F, van der Wiel SE, Ter Borg PCJ, Koch AD, Ouwendijk RJT, Slangen RME, Siersema PD, Bruno MJ; Trans.IT foundation study group. Implementation of mandatory ERCP registration in The Netherlands and compliance with European Society of Gastrointestinal Endoscopy performance measures: a multicenter database study. Endoscopy. 2022 Mar;54(3):262-267. doi: 10.1055/a-1499-7477. Epub 2021 Jun 9. PMID 34107538
- [Background] Lantinga MA, Theunissen F, Ter Borg PCJ, Bruno MJ, Ouwendijk RJT, Siersema PD; Trans.IT foundation study group. Impact of the COVID-19 pandemic on gastrointestinal endoscopy in the Netherlands: analysis of a prospective endoscopy database. Endoscopy. 2021 Feb;53(2):166-170. doi: 10.1055/a-1272-3788. Epub 2020 Oct 20. PMID 33080630
- [Background] Domagk D, Oppong KW, Aabakken L, Czako L, Gyokeres T, Manes G, Meier P, Poley JW, Ponchon T, Tringali A, Bellisario C, Minozzi S, Senore C, Bennett C, Bretthauer M, Hassan C, Kaminski MF, Dinis-Ribeiro M, Rees CJ, Spada C, Valori R, Bisschops R, Rutter MD. Performance measures for ERCP and endoscopic ultrasound: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. Endoscopy. 2018 Nov;50(11):1116-1127. doi: 10.1055/a-0749-8767. Epub 2018 Oct 19. PMID 30340220
- [Background] Johnson G, Webster G, Boskoski I, Campos S, Golder SK, Schlag C, Anderloni A, Arnelo U, Badaoui A, Bekkali N, Christodoulou D, Czako L, Fernandez Y Viesca M, Hritz I, Hucl T, Kalaitzakis E, Kylanpaa L, Nedoluzhko I, Petrone MC, Poley JW, Seicean A, Vila J, Arvanitakis M, Dinis-Ribeiro M, Ponchon T, Bisschops R. Curriculum for ERCP and endoscopic ultrasound training in Europe: European Society of Gastrointestinal Endoscopy (ESGE) Position Statement. Endoscopy. 2021 Oct;53(10):1071-1087. doi: 10.1055/a-1537-8999. Epub 2021 Jul 26. PMID 34311472
- [Background] Kochar B, Akshintala VS, Afghani E, Elmunzer BJ, Kim KJ, Lennon AM, Khashab MA, Kalloo AN, Singh VK. Incidence, severity, and mortality of post-ERCP pancreatitis: a systematic review by using randomized, controlled trials. Gastrointest Endosc. 2015 Jan;81(1):143-149.e9. doi: 10.1016/j.gie.2014.06.045. Epub 2014 Aug 1. PMID 25088919